CLINICAL TRIAL: NCT06563440
Title: Development and Evaluation of an Information Management System and Communication System for Population-wide Point-of-care Infant Sickle Cell Disease Screening
Acronym: SIMCS SCD
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Makerere University (Other)
Collaborators: Baylor College of Medicine (Other); Ministry of Health, Uganda (Other Government)
Responsible Party: Principal Investigator, College of Health Sciences, Professor Nelson K. Sewankambo, Makerere University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: MakSOMREC-2021-254
Record Dates: First submitted 2024-08-19; First posted 2024-08-20 (Actual); Last update posted 2024-08-22 (Actual); Status verified 2024-08

CONDITIONS: Sickle Cell Disease
MeSH Terms: conditions — Anemia, Sickle Cell

STUDY DESIGN:
Intervention Model Description: Cluster randomized trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- App/digital system (Experimental): Experimental Hospital/HCs will be provided with point of care test kits and smart phones loaded with airtime credit and the SCD SIMCS app. The health workers that normally provide pediatric care at the facilities will be trained in using the kits and SCD SIMCS app. Outcome measures to compare the effectiveness of SCD screening with and without the SIMCS will include proportions of accurately interpreted assay results, parents that receive counseling, infants seen for SCD care within 1 month of screening, and infants on penicillin. Variables to compute these outcome measures will be entered into cellphone eCRFs (Controls) or automatically transmitted from the SCD SIMCS App (Experimental) and retrieved from the SCD SIMCS database. Chi-squared test and contingent 95% confidence intervals and p-values will be computed to compare the proportions between SIMCS vs. non-SIMCS hospital/HCs.
  Interventions: Other: Digital app and information system
- No App/digital system (Active Comparator): Control Hospital/HCs will be provided with point of care test kits and smart phones loaded with airtime credit BUT no SCD SIMCS app. The health workers that normally provide pediatric care at the facilities will be trained in using the kits. To enable independent verification of the accuracy of interpretation of assay results, health workers will use the smart phones to take and send a photographic caption of every used point of care test strip to a designated central study phone from which they will be downloaded into a computer database. Control infants will be IDed by study number in the SCD SIMCS database.
  Interventions: Other: Digital app and information system

INTERVENTIONS:
Other: Digital app and information system — A custom digital app and information system that consists of four modules: (1) ID module - captures child's demographic and biometric data and builds a printable QR-code; (2) Assay module - captures point of care test image, interprets, and transmits results to the central ministry of health data center; (3) Education module - stores and plays back short educational videos for pre- and post-screening counseling; (4) SCD e-Passport module - entry and display of child's salient clinical information.

SUMMARY:
Although over 75% of children with sickle cell disease (SCD) are born in sub-Sahara where the disease highly contributes to under-5 mortality and causes life-long debilitation, evidence-based strategies to control SCD are not widely implemented in this region. Early detection of SCD by universal infant screening is a pillar of SCD control. Despite the affordability and move to adopt point-of-care (POC) SCD screening assays in sub-Sahara Africa, the absence of screening information management and communication systems (SIMCS) impedes standardized, systematic, coordinated, nationwide SCD screening programs. The long-term goal of the proposed research is to develop a SCD SIMCS that will enable universal SCD screening in the sub-Sahara African setting. The objective is to test and optimize a custom SCD SIMCS app and digital network to facilitate SCD screening and then evaluate its impact on access to SCD screening and care and on clinical outcomes of children with SCD in Uganda. The central hypothesis is that the SCD SIMCS will facilitate accurate and coordinated POC SCD screening that is accessible at health centers in urban and rural Uganda. The rationale is to build a custom SCD SIMCS on existing nationwide digital and health infrastructure in Uganda to standardize use of affordable POC assays at health centers nationwide. The central hypothesis will be tested by pursuing two specific aims: 1) Develop and evaluate a four-module ≥3G cell phone app for a novel SCD SIMCS (R21 Phase); 2) Evaluate the impact of the SCD SIMCS on access to screening and care and outcomes of children with SCD (R33 Phase). The investigators will pursue these aims using an innovative combination of software design and re-organization of SCD screening workflows. These include assembly of off-the-shelf software that is compatible with iOS and Android operating systems to reliably, accurately, and handily capture, interpret, transmit, and retrieve/playback information for patient's IDs, test results, salient clinical events, and education. The novel screening workflows are expected to dramatically reduce the cost and increase access to SCD screening and care. The proposed research is significant, because it will determine how to use POC SCD screening assays on a large nationwide scale. It will also enable coordination of evidence-based care and continuity of care between primary and specialist providers and longitudinally over the patient's lifetime - a critical aspect in controlling this life-long disease. The SCD SIMCS will also facilitate real time data management for research and policy for SCD control. The expected immediate outcome of this research is a SCD SIMCS that optimally functions on the digital and health infrastructure in Uganda and demonstration of its impact on access to SCD screening and care and on clinical outcomes of children with SCD. The expected long-term outcome is that the SCD SIMCS will be adopted, integrated, and scaled-up in the health systems of Uganda and other sub-Sahara Africa countries, particularly those where the POC assays have already been adopted as the national standard of SCD screening. If effective, the SCD SIMCS will have an important positive impact because it will reduce the cost of SCD screening, take screening services and evidence-based care closer to rural communities where the majority of children in sub-Sahara Africa live, and, ultimately, save millions of children from preventable and disability death.

DETAILED DESCRIPTION:
This trial builds on our multidisciplinary experience in pediatric sickle cell disease (SCD) care, mHealth platforms, and community-based research in Uganda to develop, validate, and trial a novel SCD screening information management and communication system (SCD SIMCS) that enables community-wide point-of-care (POC) SCD screening and care coordination. The SCD SIMCS network will be built on existing population-wide digital infrastructure and a Tier2 data center at the Uganda Ministry of Health (MOH) hub. The network will consist of 3 components: (1) ≥2G cell phone (patients) for short message service (SMS); (2) ≥3G cell phone (providers) for a custom Application (App) that facilitates SCD testing, patient education, and care coordination; (3) Tier2 data center (MOH hub) to receive, curate and transmit data and information in the SCD SIMCS network. The network will involve families, primary care providers (PCP), pediatric hematology specialists, and a national MOH hub for SCD screening. The purpose is to improve outcomes of children with SCD through early detection and linkage into care.

SCD is a group of inherited chronic red blood cell (RBC) disorders characterized by chronic hemolytic anemia, pain crises, and end-organ damage. SCD affects about 15 million individuals in SSA, and about 340,000 children are born with the disease annually. Only 10% of these children reach adolescence in SSA compared to almost 90% of patients that reach adulthood in high-income countries.3 Although SCD contributes about 16% of under-5 mortality in SSA, it is under-recognized because most children die of the disease without a diagnosis.

Early detection through screening is the foremost strategy in reducing SCD morbidity and mortality because it is a pre-requisite for prevention of complications using interventions such as hydroxyurea, vaccination, and health education.24 Whereas several assays for SCD screening exist, attempts to introduce them in SSA at a large scale have been futile because of the unaffordable logistics and complex workflows involved in traditional designs of infant screening programs. Transportation of samples and maintenance of sample-patient ID, transmission of test results to families and providers, pre- and post-screening counseling, referral for treatment for those diagnosed with SCD, and program evaluation are all critical steps in screening and are dependent on affordability, reliability, and integrity of information transfer between the stakeholders at each step. The investigators hypothesize that the SCD SIMCS will bridge these gaps in the screening process in Uganda and sustainably improve outcomes of children with SCD. The investigators propose the following Specific Aims to develop, validate, and trial a sustainable and error-proof mHealth system that will subsequently be adoptable and sustainable to facilitate population-wide SCD screening in Uganda:

Aim 1. To develop and evaluate a four-module ≥3G cell phone app for a novel SCD screening information management and communication system (SIMCS) (R21 Phase). The App will capture and interpret POC assays, capture and maintain a high-fidelity patient ID system, serve as a SCD e-passport interface, and facilitate SCD pre- and post- test counseling. The investigators will iteratively test the feasibility, accuracy, reproducibility, efficacy and robustness of the custom App and SCD SIMCS in our Mulago National Referral Hospital (MNRH)/Makerere University College of Health Sciences (MakCHS) Sickle Cell Program and affiliated primary health centers in Kampala. The goal is to enable a simple, error-free, reliable, and standardized SCD screening using a low-cost POC assay that can be performed across wide ranging health center levels and health worker expertise, and facilitate efficient information sharing and coordination between stakeholders.

Aim 2: To evaluate the impact of the SCD SIMCS on access to screening and care and outcomes of children with SCD (R33 Phase). Hypotheses: The SCD SIMCS will enable universal SCD screening of infants in participating communities, facilitate coordination of their clinical care, and result in reduction of morbidity and mortality due to SCD in participating communities. The investigators will perform a clustered randomized trial (CRT) of the SCD SIMCS among health centers in one urban and three rural districts of Uganda. The goal is to generate community level evidence on the impact of the SCD SIMCS to inform its adoption and expansion to a national scale in Uganda, and adaptation to other LMIC countries.

In Phase 1 the investigators will finalize creation of short videos for patient education, integrate the modules of the SCD SIMCS ≥3G cell phone App and test its integration with the Ministry of Health (MOH) Tier3 data center. The investigators will also optimize the analytics and informatics algorithms for data transmitted to the MOH data center. Reiterations of improvements and testing to optimize the design and functionalities of the App and SCD SIMCS will be made based on user feedback. Phase 1 will be conducted at Mulago National Referral Hospital and, later, piloted in a sample of health centers in the city of Kampala. In Phase 2 the investigators will conduct a Cluster Randomized Trial (CRT) involving health centers in one urban district (Kampala) and three rural districts that have established community research infrastructure; the Iganga-Mayuge Health Demographic Survey Site (IMHDSS) and Rakai Health Research Program (RHRP).

The investigators expect the proposed SCD SIMCS to reduce SCD mortality and morbidity by expanding access to screening, facilitating continuity and coordination of care, and providing real time data for national SCD policy and planning and research. Our team involves stakeholders with the mandate and resources to successfully conduct the proposed research and, most critically, to integrate and sustain the SCD SIMCS in the health system.

ELIGIBILITY:
Inclusion Criteria: A participant will be eligible for enrolment if at baseline they are an infant less than 1 year of age and presents to any of the health centers in the communities where the project will be conducted.

Exclusion Criteria: Persons 1 year or older

Max Age: 5 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 24000 (Estimated)
Dates: Start 2024-08-21 (Estimated); Primary Completion 2027-07-31 (Estimated); Study Completion 2028-07-31 (Estimated)

PRIMARY OUTCOMES:
Access to sickle cell disease screening and care | One month from screening for sickle cell disease
  Proportion of infants with sickle cell disease seen at health center within one month of diagnosis
Access to evidence-based care for sickle cell disease | One year from diagnosis of sickle cell disease
  Proportion of children under five that are diagnosed with sickle cell disease and receiving penicillin prophylaxis
Impact of a coordinated screening and treatment program | Two years from diagnosis of sickle cell disease
  Adjusted mortality rate for children with sickle cell disease

SECONDARY OUTCOMES:
Cost of sickle cell disease screening | Two years
  Financial cost per child screened
Access to evidence-based care for sickle cell disease | Two years from diagnosis of sickle cell disease
  Proportion of children with sickle cell disease on hydroxyurea therapy
Impact of a coordinated screening and treatment program | Two years
  Prevalence of complications of sickle cell disease including erythrocyte transfusion, sepsis, stroke, and growth delay

CONTACTS AND LOCATIONS:
Locations (2):
- Baylor College of Medicine, Houston, Texas, United States
- College of Health Sciences, Makerere University, Kampala, Uganda

IPD SHARING:
Plan to Share IPD: No